CLINICAL TRIAL: NCT06853405
Title: NUTRIMIND: Nutrition-based Interventions to Prevent Cognitive Decline
Brief Title: Nutrition-based Interventions to Prevent Cognitive Decline
Acronym: NUTRIMIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Saude Publica da Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NUTRIMIND_2024
Record Dates: First submitted 2025-02-27; First posted 2025-03-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Dysfunction; Cognition Disorder; Memory Disorders; Cognitive Impairment; Neurocognitive Disorders
Keywords: Healthy Aging; Dementia; Cognitive Dysfunction; Diet, Food and Nutrition; Diet, Mediterranean; Randomized Controlled Trial
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders; Memory Disorders; Neurocognitive Disorders; Dementia | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: In this parallel randomized trial, eligible participants after giving their consent will be randomly allocated (1:1) into 2-arms using a sequence generated in WinPepi® software: the intervention and the control groups. Once the randomization is completed, the principal investigator will inform the participants of their group allocation. Both groups will be assessed concurrently, and participants in one group do not cross over into the other group during the study.
Who Masked: Outcomes Assessor
Masking Description: The principal investigator will generate the randomization sequence, will inform the participants of their allocation group and will be responsible for the intervention's sessions. The assessors will not know each participants' allocation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NUTRIMIND (Experimental): The NUTRIMIND arm will be invited to receive a multidomain nutrition-based intervention to prevent cognitive decline, including lifestyle group sessions of nutrition education, daily activities to reduce physical inactivity, as well as individualized cognitive training and individualized clinical nutrition consultations. They will continue receiving the usual standard care in their healthcare unit.
  Interventions: Behavioral: Nutrition-related lifestyle group sessions; Behavioral: Cognitive training; Behavioral: Clinical nutrition consultations
- Control (No Intervention): The control arm will receive a healthy recipe cookbook and will also be invited to attend free healthy cooking workshops after the data collection phase concludes. And will continue receiving the usual standard care in their healthcare unit.

INTERVENTIONS:
Behavioral: Nutrition-related lifestyle group sessions — In person lifestyle group sessions of 180-minutes per week, directed by a nutritionist, and comprising:
  1. nutrition education session for preparing healthy meals, followed by a period of social interaction while consuming the meals prepared. Participants will be encouraged to apply the healthy cooking techniques covered in each session in their home context.
  2. daily activities to reduce physical inactivity (e.g., walking to the supermarket to buy ingredients, playing traditional games, caring for community gardening, among others).
  Arms: NUTRIMIND
Behavioral: Cognitive training — Individualized cognitive training performed remotely, at home on their own. The participants will be invited to perform cognitive training exercises at least twice a week using COGWEB®, an online platform for cognitive training. For those unable to use computer devices, similar exercises will be available in paper-and-pencil format.
  Arms: NUTRIMIND
Behavioral: Clinical nutrition consultations — A registered nutritionist will conduct individualized clinical nutrition consultations to each participant three times over the course of the study period.
  Arms: NUTRIMIND

SUMMARY:
This study intends to evaluate the feasibility and the effectiveness of an innovative and integrated nutrition-based intervention addressing key modifiable risk factors for dementia while meeting participants' preferences for nutrition-related sessions. The intervention will include lifestyle group sessions regarding nutrition education and physical activity, individualized cognitive training at home, as well as clinical nutrition consultations.

DETAILED DESCRIPTION:
The present project is a randomized controlled trial (RCT) to study the feasibility and effectiveness of a 6-month nutrition-based intervention designed to prevent cognitive decline in adults at higher risk of dementia.

Eligible individuals (n=120) recruited at primary health care centers or in the community will be randomized (1:1) into two arms: intervention and control groups.

The intervention group will be invited to participate in nutrition-based sessions of 180-minutes per week, directed by a nutritionist, to improve participants' skills in preparing healthy meals and reduce sedentary behaviours. Participants will also be asked to perform cognitive training at home and to attend individualized clinical nutrition consultations.

The control group will participate in data assessment and will receive a healthy recipes cookbook to thank for their participation. They will also receive an invitation to participate in free healthy cooking workshops, which will be offered upon the completion of the primary data collection endpoint.

Both groups will continue receiving the usual standard care in their healthcare unit.

Participants' assessments will be performed at baseline and will be repeated at the end of intervention (6 months after the beginning of the intervention). A follow-up assessment will be conducted 6 months after the intervention concludes. Adherence outcomes, as well as lifestyle, health and anthropometric data, cognitive performance, subjective memory complaints, anxiety and depression, quality of life and self-reported physical activity will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 55 to 85 years old;
* At least 4 years in the regular school system;
* Higher individual risk for dementia defined as a score ≥6 points on the Cardiovascular Risk Factors, Aging and Dementia Dementia Risk Score (CAIDE).

Exclusion Criteria:

* Montreal Cognitive Assessment (MoCA) score lower than the validated cutoff points defined as 2 standard deviations below the normative reference value for the corresponding age and education in the Portuguese population;
* Having a medical condition limiting the participation in the intervention (e.g., blindness, amputation…);
* Lack of autonomy in daily activities;
* Diagnosis of dementia or major incapacity.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Self-reported adherence to the Mediterranean Diet | Up to 6 months
  Variation of participant's self-reported adherence to the Mediterranean diet, assessed using the Mediterranean food pattern scale (MEDAS), between the baseline assessment and the end of the intervention. This scale varies from 0 (lowest adherence to the Mediterranean diet) to 14 points (highest adherence to the Mediterranean diet). A score ≥ 10 points indicates good adherence to the Mediterranean diet.
Self-reported quality of life | Up to 6 months
  Variation of participant's quality of life, assessed using the EuroQol Group scale - 5 dimensions (EQ-5D) scale, between the baseline assessment and the end of the intervention. This scale is subdivided into two subscales: a) five multiple choice questions, with five response possibilities, which produce a score that varies from 5 (best score) to 25 points (worst score); b) visual analogic scale, that varies from 0 (worst score) to 100 (best score).

SECONDARY OUTCOMES:
Self-reported memory complaints | Up to 6 months
  Variation of the self-reported memory complaints, assessed using the Subjective Memory Complaints Scale, between the baseline assessment and the end of the intervention. This scale varies from 0 (best score) to 21 points (worst score). Scores > 3 points indicate the presence of self-reported memory complaints.
Cognitive performance 1 | Up to 6 months
  Participant's cognitive performance assessed using the Montreal Cognitive Assessment, between the baseline assessment and the end of the intervention. In this scale the worst cognitive performance is equal to 0 and the best cognitive performance is equal to 30 points.
Cognitive performance 2 | Up to 6 months
  Variation of participant's cognitive performance assessed using the Portuguese version of Addenbrooke's Cognitive Examination - Revised (ACE-R), between the baseline assessment and the end of the intervention. This brief test evaluates the following cognitive subdomains: attention and orientation, memory, fluency, language and visuospatial. The test is scored from 0 to 100 points (highest possible score). Higher scores will indicate better cognitive performance.
Anxiety and depression symptoms | Up to 6 months
  Variation of the anxiety and depression scores, assessed using the Hospital Anxiety and Depression Scale (HADS), between the baseline assessment and the end of the intervention. This scale varies from 0 (best score) to 21 points (worst score).
Blood Pressure | Up to 6 months
  Variation of participant's systolic and diastolic blood pressure, between the baseline evaluation and the end of the intervention.
Body Mass Index | Up to 6 months
  Variation of participant's body mass index between the baseline assessment and the end of the intervention.
Self-reported physical activity | Up to 6 months
  Variation of participants' self-reported physical activity using the short version of the International Physical Activity Questionnaire (IPAQ), between baseline and the end of the intervention. Participants will be classified into 3 levels of physical activity: inactive, minimally active and active.
Health Literacy | Up to 6 months
  Variation of participant's health literacy Portuguese validated version of the NVS - Newest Vital Sign between baseline assessment and the end of the intervention. The NVS includes six questions regarding an ice cream nutrition label. The scores range from 0 to 6 (1 point for each correct answer): a score of 0 - 1 suggests high likelihood of limited literacy; 2 - 3 indicates the possibility of limited literacy; and 4 - 6 almost always indicates adequate literacy.
Nutrition Knowledge on Mediterranean Diet for Cardiovascular Disease | Up to 6 months
  Variation of participants' nutrition knowledge about Mediterranean Diet and its health benefits between baseline assessment and the end of the intervention. The nutrition knowledge will be assessed using a 20-item tool, the Mediterranean Diet Nutrition Knowledge Questionnaire (Med-NKQ). In total, the tool score range from 0 to 42, with a higher score indicating greater knowledge.
Adherence to each intervention | Up to 6 months
  Proportion of adherence to each intervention, calculated as the number of sessions attended divided by the total number of sessions implemented.
Dropout | Up to 6 months
  Proportion of participants who dropped out of the study, calculated as the number of participants who dropped out after attending at least one session divided by the total number of participants who attended at least one session.
Time of follow-up | Up to 6 months
  Number of days between the first and the last session attended by the participant.
Implemented sessions | Up to 6 months
  Proportion of sessions implemented, calculated as the number of sessions that the research team was able to implement divided by the total number of sessions planned.
Complete assessment of participants | Up to 12 months
  For each study outcome, proportion of participants with complete information, calculated at baseline and different moments of follow-up, as the number of participants with complete information divided by the total number of participants evaluated.

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Instituto de Saúde Pública da Universidade do Porto, Porto, Portugal
  - Faculty of Nutrition and Food Sciences, University of Porto, Porto

IPD SHARING:
Plan to Share IPD: Undecided